CLINICAL TRIAL: NCT06317857
Title: Clinical Performance of an Alkasite-based Restorative Material Versus Highly Viscous Glass Ionomer in Occlusal Cavities After 18 Months: A Randomized Clinical Trial
Brief Title: Clinical Performance of an Alkasite-based Restorative Material
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Tarek Mohamed Tawfik Alagamawy, Doctor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14422021443228
Record Dates: First submitted 2024-03-01; First posted 2024-03-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Caries, Dental
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Centio Forte (Ivoclar). (Experimental): A new class of bioactive "alkasite" restorative materials has been released in the market. They're composed of three main filler types: salinized inert barium aluminium silicate glass, calcium barium aluminium fluorosilicate glass similar to glass-ionomers, and calcium fluorosilicate glass or "alkasite" glass. Cention N (Ivoclar Vivadent) was the first available material in the material in the form of powder/liquid, later on, Cention forte was released which is the modified capsulated form with a special adhesive system Marovic et al. (2022).
  Cention has the ability to remineralize hard dental tissues through calcium and fluoride release and can also neutralize bacterial acids through hydroxide ions release Par et al. (2020).
  Interventions: Other: Centio Forte
- Highly viscous glass ionomer (Active Comparator): Glass-ionomer restorations (GI) are widely used in restorative dentistry. One of their advantages is their chemical adhesion to tooth structure. They also possess a fluoride-releasing property and biocompatibility. Although GIs are commonly used, they have some disadvantages. The most intractable problem with the conventional GIs is probably their lack of strength and toughness. In order to improve the mechanical properties of conventional GICs, reinforced GIs were developed. These reinforced GIs or now commonly known as highly viscous GIs provide improved mechanical properties and wear resistance, easier application allowing their use in posterior stress bearing cavity preparations Bakhadher et al.
  (2019).
  Interventions: Other: Centio Forte

INTERVENTIONS:
Other: Centio Forte — A new Alkasite material has been introduced with superior strength and bioactive ion release where it is considered the new alternative to amalgam.

SUMMARY:
The evolution of restorative dental materials and technology has enabled the use of tooth-colored restorative materials in dental restorations, with all dentists hoping for the presence of materials that combine biocompatible qualities and aesthetics . Although resin composite materials' mechanical and aesthetic properties have greatly improved over the past 20 years, research is currently on to find ways to prevent secondary caries from forming beneath and at the margins of restorations. In order to circumvent these problems, there is a growing tendency towards the use of resin-based bioactive and remineralizing restorative materials to strengthen and lengthen the lifespan of bonded dental restorations.

DETAILED DESCRIPTION:
The evolution of restorative dental materials and technology has enabled the use of tooth-colored restorative materials in dental restorations, with all dentists hoping for the presence of materials that combine biocompatible qualities and aesthetics . Although resin composite materials' mechanical and aesthetic properties have greatly improved over the past 20 years, research is currently on to find ways to prevent secondary caries from forming beneath and at the margins of restorations. In order to circumvent these problems, there is a growing tendency towards the use of resin-based bioactive and remineralizing restorative materials to strengthen and lengthen the lifespan of bonded dental restorations.Glass ionomer is one of the most commonly used materials in dental restorations. One of the most important properties of GICs is their ability to release fluoride and recharge. Other reasons for GIC's widespread use in the dental field are its beneficial properties such as adhesion to tooth structure, equivalent coefficient of thermal expansion of teeth, and excellent biocompatibility. However, they have disadvantages such as severe wear, high solubility, poor mechanical properties, and limited occlusal force resistance. Today's generation GICs have tried to address these disadvantages by incorporating a fast setting reinforced glass ionomer that should offer protection during the early maturation process and enhance strength and surface hardness. It has been improved by changes in the ratio of powder to liquid, particle size and dispersion. As a result, highly viscous glass ionomer (HVGIC) is available on the market. In the last few years, we have seen the introduction of a glass ionomer encapsulated with high mechanical properties as claimed by the manufacturer. The GIC, which is characterized by its rapid setting and high viscosity, could serve as an alternative to amalgam and composite restorations in cavities of class I and II for permanent teeth.

For decades, dentists have been looking for a material that is affordable, fluoride releasing, easy to apply, strong, and aesthetically pleasing. A novel bioactive, alkasite material has been introduced enabling quick and efficient minimally invasive treatment. . It is a self-curing radiopaque material for direct treatment of anterior and posterior cavities. It is claimed as a tooth coloured, bioactive, durable material to be rendered as the new alternative to amalgam for permanent Class I and II restorations. It also promotes remineralization and prevents demineralization with an advanced ion-releasing system. When the pH drops because of the growth of the cariogenic bacteria, it releases hydroxide ions to help restore the pH balance. Hydroxide ions help to prevent tooth structure from being demineralized. The fluoride and calcium ions released help remineralize the tooth structure and prevent secondary caries.

ELIGIBILITY:
Inclusion Criteria:

* • Patients with carious occlusal lesions with underlying dark shadow in posterior teeth (lower first molar) with ICDAS score 4.

  * Patients with at least 20 teeth under occlusion.
  * Age: 16-55 years.
  * Co-operative patients approving to participate in the trial.

Exclusion Criteria:

* • Patients younger than 16 years old or older than 55 years old.

  * Extensive occlusal lesions.
  * Teeth with signs and symptoms of irreversible pulpitis or pulp necrosis.
  * Teeth supporting removable prostheses, or orthodontic appliances.
  * Candidates with parafunction or bruxism.
  * Candidates with systemic diseases or disabilities that may affect participation.
  * Drug-induced xerostomia.
  * Heavy smoking.
  * Pregnancy.
  * Lack of compliance.

Ages: 16 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 68 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Retention success rate % with modified USPH criteria | 18 months with; T0=Baseline, T1= 6 months follow up, T2=12 months follow up and T3= 18 months follow up.
  retention of the restoration, with USPH criteria

SECONDARY OUTCOMES:
Marginal adaptation with modified USPH criteria marginal discolouration, recurrent caries, anatomic form and postoperative sensitivity. | 18 months with; T0=Baseline, T1= 6 months follow up, T2=12 months follow up and T3= 18 months follow up.
  marginal integrity of the restoration with USPH criteria
Postoperative sensitivity | 18 months with; T0=Baseline, T1= 6 months follow up, T2=12 months follow up and T3= 18 months follow up.
  Degree of post operative sensitivity with USPH criteria

IPD SHARING:
Plan to Share IPD: No